CLINICAL TRIAL: NCT05211791
Title: Comparison Between Thoracic Epidural Anaesthesia, Erector Spinae Block and Paravertebral Block During Single-lung Ventilation for Lung Resection in Lateral Decubitus Position: A Prospective Randomized Study
Brief Title: TEA, ESB and Paravertebral Block During Single-lung Ventilation for Lung Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Egypt Cancer Institute (Other)
Responsible Party: Principal Investigator, Alaa Ali M. Elzohry, Lecturer of Anesthesia, ICU and Pain Relief, South Egypt Cancer Institute, Assiut University, Egypt, South Egypt Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TEA in single lung ventilation
Record Dates: First submitted 2022-01-02; First posted 2022-01-27 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Lung Diseases; Pain, Acute
MeSH Terms: conditions — Lung Diseases; Acute Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group TEA (Active Comparator): insertion of Thoracic epidural anesthesia plus GA with lung isolation using suitable size double lumen tube at level T6
  Interventions: Procedure: Thoracic epidural anesthesia
- Group ESB (Active Comparator): U/S guided erector spinae block anesthesia using 15 ml local anesthesia plus GA with lung isolation using a suitable size double-lumen tube
  Interventions: Procedure: erector spinae block
- Group PVB (Active Comparator): U/S guided paravertebral block anesthesia using 15 ml local anesthesia as total volume plus GA with lung isolation using suitable size double lumen tube
  Interventions: Procedure: paravertebral block anesthesia

INTERVENTIONS:
Procedure: erector spinae block — Ultrasound-guided insertion of different analgesic procedures as paravertebral block anesthesia and paravertebral block anesthesia
  Arms: Group ESB
Procedure: paravertebral block anesthesia — Ultrasound-guided insertion of different analgesic procedures as paravertebral block anesthesia and paravertebral block anesthesia
  Arms: Group PVB
Procedure: Thoracic epidural anesthesia — insertion of Thoracic epidural catheter for anesthesia analgesia at level of T6
  Arms: Group TEA

SUMMARY:
Thoracotomy operations are known to be painful surgical procedures, so providing effective intraoperative and postoperative analgesia is so important for all anaesthesiologists. Ineffective pain management interferes with deep breathing, coughing, and remobilization resulting in atelectasis and pneumonia.

Ultrasound-guided ESP block is a myofascial plane block that provides analgesia for thoracic or abdominal segmental innervation depending on the level of the injection site. Thoracic epidural analgesia (TEA) is considered the gold standard analgesic technique for thoracic surgeries. But the invasiveness of this technique, the rare but serious neurologic complications and the failure rates up to 30% are the disadvantages of epidural analgesia

DETAILED DESCRIPTION:
The aim of this study is to compare the effect of different blocks as TEA, erector spinae block or paravertebral block on improving peri-operative analgesia and post-operative outcome in pulmonary resection in adult patients.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 to 70 years old for elective lung resection. with American Society of Anesthesiology physical status (ASA-PS) I-III

Exclusion Criteria:

* Total pneumonectomy
* Hepatic or renal dysfunction.
* contraindications for epidural anesthesia as Coagulopathy and neurological and spinal deficits.
* emergency cases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-06-10 (Estimated); Study Completion 2023-10-20 (Estimated)

PRIMARY OUTCOMES:
peri-operative analgesia | up to 48 hours postoperative
  Visual Analogue score (resting and during cough) from 0 (no pain) to 10 (worst pain pain measurement

CONTACTS AND LOCATIONS:
Overall Officials: Alaa A Elzohry, Principal Investigator — Lecturer of Anesthesia , ICU and pain management
Locations (1):
- South Egypt Cancer Institute, Assiut University, Arab Republic of Egypt, Asyut, Egypt